CLINICAL TRIAL: NCT01532531
Title: The Effects of Collateral Meridian Therapy for Knee Osteoarthritis Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Huei-Chi Horng, MD, Principal Investigator, Taichung Armed Forces General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TC98-2
Record Dates: First submitted 2012-02-07; First posted 2012-02-14 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Knee Osteoarthritis; Pain
Keywords: Collateral Meridian Therapy; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collateral Meridian Therapy (Experimental): The CMT group patients received, according to the CMT protocol described previously, CMT at the selected points with the CMT Electrotherapy Stimulator ("GEMORE" Multi-Function Electrotherapy Stimulator; GM390TE, GEMORE Co Ltd, Taiwan) to treat the affected OA knee. The 6-minute treatment (electrotherapy was set at 40 Hz biphasic and 30 mA) comprises reduction and enhancement procedures on the specific points. Each patient received CMT twice per week for three weeks during the study.
  Interventions: Device: "GEMORE" Multi-Function Electrotherapy Stimulator
- Control (CT) group (No Intervention): Patients in the CT group received electronic lead-patches applied on the treatment points, which was identical to what the CMT patients received, also for 6 minutes, though no electric stimulation was applied.

INTERVENTIONS:
Device: "GEMORE" Multi-Function Electrotherapy Stimulator — The Collateral Meridian Therapy (CMT) group patients received, according to the CMT protocol described previously (5), CMT at the selected points with the CMT Electrotherapy Stimulator ("GEMORE" Multi-Function Electrotherapy Stimulator; GM390TE, GEMORE Co Ltd, Taiwan) to treat the affected OA knee. The 6-minute treatment (electrotherapy was set at 40 Hz biphasic and 30 mA) comprises reduction and enhancement procedures on the specific points. Each patient received CMT twice per week for three weeks during the study.
  Arms: Collateral Meridian Therapy

SUMMARY:
Collateral meridian therapy (CMT) is a recently developed technique according to traditional Chinese medicine (TCM) experiences, differing from traditional Chinese acupuncture in numerous manners. CMT involves the manipulation of a distant non-painful collateral meridian, thereby facilitating the dissipation of pain. The technique avoids direct stimulation of the involved meridian, which enhances patient tolerability and prevents further injury to the disease and painful areas. Numerous clinical cases have reported the effectiveness of CMT in pain management. This study tests whether CMT is effective for treating knee OA pain and functional recovery.

DETAILED DESCRIPTION:
Knee OA patients aged 60 years or older were recruited from the orthopedic clinic of Taichung Armed Force General Hospital, Taichung, Taiwan. All the patients had been clinically and radiologically diagnosed with knee OA according to the criteria of the American College of Rheumatology and Lawrence radiographic changes in the tibiofemoral joint by using a visual analogue scale (VAS) pain score higher than 30 mm on a 100-mm scale over the medial side of the knee while walking. Individuals who had undergone total knee arthroplasty, exhibited uncontrolled hypertension, had a history of cardiovascular disease, or suffered from neurological disorders that affected lower extremity functions were excluded from the study. Patients who received conflicting or ongoing interventions such as acupuncture, hyaluronan injections, intra-articular corticosteroid, and transcutaneous electrical nerve stimulation and thermotherapy were also excluded. Patients under drug treatment were included if no changes in medication had occurred, and the dosages had been administered for one month or longer. Oral paracetamol or non-steroidal anti-inflammatory drugs (NSAIDs) were permitted as rescue pain medications for the duration of the study. Rescue pain medications or any change in medicines and dosages were recorded. This study was approved by the IRB of Tri-Service General Hospital, Taipei, Taiwan and written informed consents were obtained from the enrolled participants. According to the sealed envelop method, the enrolled patients were randomly allocated to the control group or CMT group.

Treatment CMT group The CMT group patients received, according to the CMT protocol described previously, CMT at the selected points with the CMT Electrotherapy Stimulator ("GEMORE" Multi-Function Electrotherapy Stimulator; GM390TE, GEMORE Co Ltd, Taiwan) to treat the affected OA knee. In brief, knee OA mostly induced knee pain at the medial side, the corresponding disease meridian of OA is AxI/3, the first yin meridian (AxI) over knee region ("3") on the medial aspect of the lower extremity (the spleen meridian in TCA). A reduction technique, to remove the obstructed overflowed Qi, was performed by treating the point "3" on the ipsilateral third yang meridian (TyIII) over the dorsal aspect of the upper extremity (TyIII/3:3), which corresponded to Tze Cheng (SI7) on the small intestine meridian in TCA; the aspect shares the same control C-point (the first "3" ) and F-point (the second "3") to divert the obstructed Qi from obstructed diseased meridian to the healthy one; the C-point is used to link the diseased meridian to the treatment healthy meridian; manipulating the F-point is for the treatment/removal of the disease/pain symptom. An enhancement technique was performed by treating contralateral meridian "Ax II/2:(3)," which represents treating "2" as the C-point and "3" as the F-point, and a number in parentheses signifies usage of enhancement technique on the contralateral second yin meridian of the medial aspect of the lower extremity (corresponding to San Yin Jiao (SP6) and Lou Ku (SP7), respectively, on the liver meridian in TCA). The 6-minute treatment (electrotherapy was set at 40 Hz biphasic and 30 mA) comprises reduction and enhancement procedures on the specific points (figures 1 and 2). Each patient received CMT twice per week for three weeks during the study.

Control (CT) group The patients in the CT group received electronic lead-patches applied on the treatment points, which was identical to what the CMT group received, also for 6 minutes, though no electric stimulation was applied.

Evaluation of outcomes Primary outcome measures were: (1) pain intensity at activity, quantified with a 100 mm VAS and (2) pain disability measured with the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC, 0-96 points). The WOMAC is a disease-specific measure of pain, stiffness, and physical function for individuals with knee OA. The WOMAC comprises 5 items related to pain, 2 items related to stiffness, and 17 items related to physical function. Each item is scored on a 5-point Likert scale (0-4). The reliability and validity of WOMAC scores have been established. The VAS and WOMAC scores were measured immediately by independent staff before the first treatment, and subsequently at one, two, three weeks, and three months after the first treatment.

Statistical analysis Patients were excluded from analysis if they were not present for the follow-up, or the outcomes were not assessed. The Mann-Whitney test was employed to analyze differences between the VAS and WOMAC scores of the two groups. SPSS software for Windows was used for statistical analysis. All the data are presented as means (±SD). The data with P values less than 0.05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA patients aged 60 years or older
* Visual analogue scale (VAS) pain score higher than 30 mm on a 100-mm scale over the medial side of the knee while walking

Exclusion Criteria:

* Individuals who had undergone total knee arthroplasty, exhibited uncontrolled hypertension, had a history of cardiovascular disease, or suffered from neurological disorders that affected lower extremity functions were excluded from the study.
* Patients who received conflicting or ongoing interventions such as acupuncture, hyaluronan injections, intra-articular corticosteroid, and transcutaneous electrical nerve stimulation and thermotherapy were also excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index, visual analogue scale | 3 months
  ain intensity at activity, quantified with a 100 mm VAS and pain disability measured with the Western Ontario and McMasters Universities Osteoarthritis Index. The VAS and WOMAC scores were measured immediately by independent staff before the first treatment, and subsequently at one, two, three weeks, and three months after the first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Shung Wong, PhD, Study Director — Cathay General Hospital
Locations (1):
- Taichung Armed Forces General Hospital, Taichung, Taiwan